CLINICAL TRIAL: NCT01686802
Title: Oral Morphine Versus Ibuprofen for Post-operative Pain Management in Children: a Randomized Controlled Study
Brief Title: Post-operative Oral Morphine Versus Ibuprofen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Naveen Poonai, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 102923
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Post-operative Pain
Keywords: oral morphine; ibuprofen; post-operative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ibuprofen (Active Comparator): ibuprofen 10 mg/kg (max 600 mg) every 6 hours as needed for pain (maximum 8 doses) from the time the patient is discharged from hospital as deemed by the physician to a maximum of 48 hours.
  Interventions: Drug: Ibuprofen
- oral morphine (Active Comparator): oral morphine 0.5 mg/kg (max 20 mg) every 6 hours as needed for pain (maximum 8 doses) from the time the patient is discharged from hospital as deemed by the physician to a maximum of 48 hours.
  Interventions: Drug: oral morphine

INTERVENTIONS:
Drug: oral morphine
  Arms: oral morphine
Drug: Ibuprofen
  Arms: ibuprofen

SUMMARY:
Children 5-17 years of age who have undergo orthopedic day surgical procedures for definitive management of fractures, tendon release, etc. will be randomized to receive either ibuprofen or oral morphine as needed for pain relief for 48 hours post-operatively at home. Pain will be assessed using the self-report Faces pain scale revised (FPS-R). We hypothesize that oral morphine will result in significantly lower pain scores on the Faces Pain Scale Revised (FPS-R) compared to ibuprofen. It is hoped that the results of this trial will create a new option for post-operative pain management in children.

ELIGIBILITY:
Inclusion Criteria:

* all children aged 5-17 years who undergo an elective orthopedic or fracture-related surgical procedure at the Children's Hospital in London, Ontario and have a same-day discharge.

Exclusion Criteria:

* known hypersensitivity to either ibuprofen or morphine
* chronic users of NSAIDS or opioids
* cognitive impairment
* poor English fluency
* pregnancy
* acute or chronic renal insufficiency
* bleeding disorder
* obstructive sleep apnea

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 132 (Actual)
Dates: Start 2012-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in faces pain score pre and post intervention | 48 hours from the time of discharge from hospital.

SECONDARY OUTCOMES:
Change in faces pain score pre and post intervention | 48 hours from the time of discharge from hospital
  Second to eighth doses of intervention
Adverse effects | 96 hours from first dose of intervention
Number of participants requiring acetaminophen for breakthrough pain | 48 hours from first dose of intervention
Unscheduled visits to a health care provider for pain | 96 hours from first dose of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Naveen Poonai, MSc MD FRCPC, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Science Center, London, Ontario, Canada

REFERENCES:
- [Derived] Poonai N, Datoo N, Ali S, Cashin M, Drendel AL, Zhu R, Lepore N, Greff M, Rieder M, Bartley D. Oral morphine versus ibuprofen administered at home for postoperative orthopedic pain in children: a randomized controlled trial. CMAJ. 2017 Oct 10;189(40):E1252-E1258. doi: 10.1503/cmaj.170017. PMID 29018084